CLINICAL TRIAL: NCT03766152
Title: Audiological Benefit and Improved Quality of Life With Two Bone Conduction Systems: ADHEAR vs. Bonebridge in Experienced Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dominik Riss (Other)
Responsible Party: Sponsor-Investigator, Dominik Riss, Assoc. Prof PD Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1757/2018
Record Dates: First submitted 2018-11-16; First posted 2018-12-06 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Bone Conduction Deafness; Hearing Loss, Conductive
Keywords: Hearing aid
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adhear (Other): Patients will be fitted with an adhesive bone conduction device for three weeks
  Interventions: Device: Adhesive bone conduction hearing aid (ADHEAR - Med El)

INTERVENTIONS:
Device: Adhesive bone conduction hearing aid (ADHEAR - Med El) — Patients are asked to wear an adhesive bone conduction hearing device which is attached to the mastoid with an adhesive adapter

SUMMARY:
Patients implanted with a Bonebridge will be asked to be part of the study. The study subjects are enrolled into the study according to inclusion criteria.

Patients will be asked to wear an adhesive bone conduction device an adapt to it for 30-60 min. After this time period patients will be asked to use the adhesive device instead of the Bonebridge for 3 weeks. Audiologic Tests and quality of life questionnaires will be assessed at the beginning of the study and at the end of three weeks.

DETAILED DESCRIPTION:
Phase 1 Patients will be fitted with an adhesive bone conduction device and asked to fill out two questionnaires. They will then wear the device for 30-60 minutes and decide if they want to wear the device for the remaining study time of three weeks. Patients who do not have sufficient benefit from the device or do not feel comfortable with it do not enter the second study period of wearing the device for three weeks. Patients will be asked to comment on their experiences after 30 to 60 minutes explaining why they do not want to enter the second part of the study if they feel comfortable sharing this information. Phase 2 Patients, in the second study period, will be asked to wear the hearing device as long as comfortable to them every day and mark time of device usage, battery life, changes of the adhesive adapter, sound quality and comfort related remarks in a diary. After three weeks patients will return to the outpatient ́s department for an audiological assessment and a second set of quality of hearing and quality of life questionnaire.

No patients will be implanted with a Bonebridge as part of the study.

Audiologic testing consists of sound field audiometry, Freiburg monosyllables test and Oldenburg sentence test.

Questionnaires consist of the AQol-8D and the SSQ-12

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a Bonebridge device and are active users
* Unilateral and/or bilateral conductive hearing loss (CHL)
* Subjects aged 13 years or older
* Capable of the German language
* Willingness and ability to perform all tests required for the study
* Signed, and dated informed consent before the start of any study specific procedure

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patient is intolerant of the materials as described by Manufacturer's IFU
* Patient presents with a skin or scalp condition that may preclude the attachment of the adhesive adapter.
* Patient cannot perform the audiological tests or is unable to fill out the questionnaires.
* Patient presents with retrocochlear, or central auditory disorder.
* any physical, psychological, or emotional disorder that would interfere with the ability to perform on test and rehabilitation procedures

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Average functional hearing gain | 3 weeks
  The primary endpoint of the study is the average functional hearing gain evaluated by the free field audiometry (at 4 different frequencies) using the bone conduction device compared to the unaided situation. To compare the two hearing devices the following primary endpoint measure will be calculated: Δmean= {(Average functional hearing gain with Bonebridge - Average functional hearing gain with ADHEAR at timepoint T1 (=Δ1)) + (Average functional hearing gain with Bonebridge - Average functional hearing gain with ADHEAR at timepoint T2 (=Δ2))} divided by two. Measuring both hearing devices at both timepoints and using the mean difference (Δmean) enables adjustment for a possible underlying customization effect.

SECONDARY OUTCOMES:
AQoL-8D (quality of life) | 3 weeks
  Will be measured by comparing Quality of Life as assessed with AQoL - 8D at the beginning of the study and the end of the study (The result of the AQoL-8D is a number)
Quality of hearing | 3 weeks
  Quality of hearing as assessed with the SSQ 12 questionnaire will be compared at the beginning of the study to the results after the three weeks with the adhesive device.
  The results of the SSQ-12 is a number
Word recognition score | 3 weeks
  Further secondary outcomes will be assessed by comparing the results of the word recognition test in the aided condition once with the implanted device (Bonebridge) in comparison to the adhesive device (ADHEAR). Word recognition is measured in percent at two different noise levels
Sentence test | 3 weeks
  Further secondary outcomes will be assessed by comparing the results of the sentence test in the aided condition once with the implanted device (Bonebridge) in comparison to the adhesive device (ADHEAR). Sentence test results are measured as percent at a certain volume level (dB).

CONTACTS AND LOCATIONS:
Locations (1):
- MUW, AKH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No